CLINICAL TRIAL: NCT05593913
Title: A Single-center, Retrospective Study to Evaluate the Clinical Performance of Artificial Intelligence Medical Assisted Diagnostic Software (VeriSee AMD) for Screening of Age-Related Macular Degeneration
Brief Title: Clinical Evaluation of VeriSee AMD in Screening for Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Acer Medical Inc. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AHCI21001
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-04

CONDITIONS: Macular Degeneration, Age Related; Maculopathy, Age Related
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study is designed to evaluate the clinical performance of VeriSee AMD for potential age-related macular degeneration (AMD) screening from color fundus photography images. The sensitivity and specificity of VeriSee AMD's automated image analysis for screening AMD will be determined through the comparison with the gold standard, which is the judgment of AMD by the ophthalmologists.

DETAILED DESCRIPTION:
This is a retrospective, single-center, observational study to assess the clinical performance of VeriSee AMD in screening for potential age-related macular degeneration (AMD).

Potential subjects with images of color fundus photography will be selected for eligibility, and then the ophthalmologist further confirms the images with legible quality. Three independent ophthalmologists (or evaluators) having more than 6 years of experience in retina will evaluate AMD from the color fundus photography images with different sequences of images independently. These three evaluators are different from the ophthalmologist who is responsible for deciding subject's eligibility. The evaluators determine the severity of AMD based on the four-level scale which is the AMD Severity Scale stated in Age-Related Eye Disease Study (AREDS) Report No. 6. Before the study, the training section is necessary to ensure the consensus of the AMD severity grading among three evaluators. The severity determined by the majority of the grade the three evaluators gave is considered the gold/reference standard in this study. Therefore, level 1 and level 2 are classified as non-mtl3AMD, while level 3 and advanced AMD (level 4) are classified as mtl3AMD. The clinical performance displayed as sensitivity and specificity will be determined by comparing the AMD results between VeriSee AMD and the gold standard.

VeriSee AMD is intended to screen AMD from the images taken by color fundus photography, which can assist the physicians to assess whether further examination for retinopathy by the ophthalmologist is needed. The screening result of AMD will be non-mtl3AMD or mtl3AMD for the physicians' reference and does not intend to diagnose AMD, detect concomitant diseases, or treat AMD.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age ≥ 50 years old
* Subject with image taken by color fundus photography that meet the following requirement:

  1. The resolution of image is 271x271 pixels or higher;
  2. The angle view of image is 45 or 50 degree.
* Subject's image includes macula as judged by the ophthalmologist.

Exclusion Criteria:

* The color fundus photography image previously used by VeriSee AMD during the development process and pre-clinical test
* The macula or other part in the image of color fundus photography is unclear to determine the disease condition as judged by the ophthalmologist.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People fifty years of age or older have color fundus photography images.
Sampling Method: Probability Sample
Enrollment: 986 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: The 986 subjects from the intended population, having at least one qualified color fundus photography image determined by the ophthalmologist, were enrolled in this study. A total of 986 color fundus photography images from all enrolled subjects were in use for effectiveness analysis.
Period: Overall Study
Arm/Group | Test Group
Started | 986
Completed | 947
Not Completed | 39
Not completed — Insufficient image quality | 39

BASELINE CHARACTERISTICS:
Population: Intended Use Population
Groups:
- Test Group: The 986 subjects from the intended patient population, having at least one qualified color fundus photography image determined by the ophthalmologist, enrolled in this study. A total of 986 color fundus photography images from all enrolled subjects were in use for effectiveness analysis.
Arm/Group | Test Group
Number analyzed (Participants) | 986
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 403
  Male | 583
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 986

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: To evaluate the clinical performance of VeriSee AMD by determining the sensitivity.
  Sensitivity = 100% x TP/(TP+FN)
Time Frame: 1 day
Population: Of 986 subjects enrolled, VeriSee AMD judged the images of 39 subjects (3.96%) as with insufficient image quality.
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Test Group: Intended Use Population
Arm/Group | Test Group
Number analyzed (Participants) | 947
percent | 90 [85.05 to 93.67]

2. Primary Outcome: Specificity
Description: To evaluate the clinical performance of VeriSee AMD by determining the Specificity.
  Specificity = 100% x TN/(TN+FP)
Time Frame: 1 day
Population: Of 986 subjects enrolled, VeriSee AMD judged the images of 39 subjects (3.96%) as insufficient image quality.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Test Group
Number analyzed (Participants) | 947
percent | 96.5 [94.88 to 97.69]

3. Secondary Outcome: Positive Predictive Values (PPV)
Description: To evaluate the clinical performance of VeriSee AMD by determining the positive predictive values (PPV).
  Positive predictive value (PPV) =100% x TP/(TP+FP)
Time Frame: 1 day
Population: Of 986 subjects enrolled, VeriSee AMD judged the images of 39 subjects (3.96%) as with insufficient image quality.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Test Group
Number analyzed (Participants) | 947
percent | 87.9 [82.71 to 91.91]

4. Secondary Outcome: Negative Predictive Values (NPV)
Description: To evaluate the clinical performance of VeriSee AMD by determining the negative predictive values (NPV).
  Negative predictive value (NPV) = 100% x TN/(FN+TN)
Time Frame: 1 day
Population: Of 986 subjects enrolled, VeriSee AMD judged the images of 39 subjects (3.96%) as with insufficient image quality.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Test Group
Number analyzed (Participants) | 947
percent | 97.1 [95.65 to 98.22]

5. Secondary Outcome: The Percentage of Subjects' Images With Insufficient Quality as Judged by VeriSee AMD
Description: The percentage of the images with insufficient quality as determined by VeriSee AMD will be presented.
Time Frame: 1 day
Population: The enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group
Number analyzed (Participants) | 986
Participants | 39

ADVERSE EVENTS:
Time Frame: This is a retrospective study and it is not necessary to collect adverse event data.
Description: This is a retrospective study and it is not necessary to collect adverse event data.
Arm/Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT05593913/Prot_000.pdf